CLINICAL TRIAL: NCT05650515
Title: The Development of a Technology-based Exercise Program for Older Adults Based on the Opinions of Older Adults and Geriatric Experts
Brief Title: A Technology-based Exercise Program for Older Adults
Acronym: Work-Oud
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PXL University College (Other)
Responsible Party: Principal Investigator, Els Knippenberg, Investigator, PXL University College
Other Study IDs: WOUD
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Older Adults; Exercise; Mobile Application
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experts: A panel of experts in the geriatric field consisting of older adults (65+ years) as well as experts (geriatric rehabilitation/medicine/research)
  Interventions: Other: Co-creation

INTERVENTIONS:
Other: Co-creation — The development of a technology-based exercise intervention based on ideas of older adults and experts in the field of geriatric rehabilitation/research/medicine

SUMMARY:
This intervention aimed to collect relevant information for the development of a technology-based exercise application. This information-collection is based on the opinions of older adults (65+ years) as well as experts from the field of geriatric rehabilitation/medicine/research.

DETAILED DESCRIPTION:
This intervention aimed to collect relevant information for the development of a technology-based exercise application. This information-collection is based on the opinions of older adults (65+ years) as well as experts from the field of geriatric rehabilitation/medicine/research.

The exercise application will be specifically designed for older adults:

* exercises targeted at endurance, strength, balance, coordination and flexibility
* importance of motivational aspects to motivate older adults to continue the program on the long term

Information that is aimed to be collected is related to a variety of aspects of the exercise application such as 1) information/education regarding the importance (health benefits) of exercise 2) design of the exercise application 3) technological aspect of the exercise application 4) motivational aspect of the exercise application

ELIGIBILITY:
Inclusion Criteria:

* Interested to contribute to the development of a technolgy-based exercise program specifically developed for older adults
* Interested to think about aspects such as "How to motivate older adults to exercise?" "Which information regarding exercise/health is relevant for older adults to motivate them to continue an exercise program?"

Exclusion Criteria:

* No interest in exercise for older adults

Ages: 65 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: Older adults (65 years or older) who have interesting/creative opinions/ideas regarding exercise (specifically for older adults), technology, health.
  Experts (no age limits) from the field of geriatric rehabilitation/research/medicine who have interesting opinions regarding exercise, technology, health specifically targeted at older adults.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Educational aspects of the exercise application | 2 days
  The collection of information from the experts and older adults regarding the educational aspect of the exercise application e.g. which educational information has te be included in the application, how? (e.g via email,...), when? (e.g. which at which time of the day)
Exercise aspect of the exercise application | 2 days
  The collection of information from the experts and older adults regarding the exercise aspect of the exercise application e.g. which exercises? which exercise equipment? Individual exercises or group exercises? With music?
Technological aspect of the exercise application | 2 days
  The collection of information from the experts and older adults regarding the technological aspect of the exercise application e.g. log in? password? kind of mobile device? which information would you like to share to complete your personal profile? GDPR aspects?
Motivational aspect of the exercise application | 2 days
  The collection of information from the experts and older adults regarding the motivational aspect of the exercise application e.g. how to motivate older adults to continue the program (and reach personal goals) on the long term? Social component of exercise (exercise in group?)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Daniëls, MSc, Principal Investigator — PXL University College
Locations (1):
- PXL University College, Hasselt, Limburg, Belgium

REFERENCES:
- [Derived] Daniels K, Vonck S, Robijns J, Quadflieg K, Bergs J, Spooren A, Hansen D, Bonnechere B. Exploring the Feasibility of a 5-Week mHealth Intervention to Enhance Physical Activity and an Active, Healthy Lifestyle in Community-Dwelling Older Adults: Mixed Methods Study. JMIR Aging. 2025 Jan 27;8:e63348. doi: 10.2196/63348. PMID 39869906
- [Derived] Daniels K, Lemmens R, Knippenberg E, Marinus N, Vonck S, Baerts J, Bergs J, Spooren A, Hansen D, Bonnechere B. Promoting physical activity and a healthy active lifestyle in community-dwelling older adults: a design thinking approach for the development of a mobile health application. Front Public Health. 2023 Nov 29;11:1280941. doi: 10.3389/fpubh.2023.1280941. eCollection 2023. PMID 38106904